## Official title:Safety and Effectiveness of Early Feeding After Bowel

### **Anastomosis in Neonates or Infants**

NCT: 04464057(This study was registered on Clinical Trials. gov)

## Primary Completion Date: 2022-12-09

A multi-center cohort was established in August 2020, and 941 case records were uploaded to http://212.64.50.165 at discharge from hospital.

## The 1st part:Safety and Effectiveness of Early Feeding After Bowel

## Anastomosis in upper, middle and lower intestinal events

#### Absract:

**Purpose** In order to prevent postoperative complications, delayed oral feeding(DOF) was still a common model of care following pediatric intestinal anastomosis surgery; however, early oral feeding(EOF) has been proven to be safe and effective in reducing the incidence of complications and fast recovery after some pediatric intestinal anastomosis. Unfortunately, evidence for initiating EOF after intestinal anastomosis in infants is insufficient. Hence, this study was primarily designed to evaluate the safety and efficacy of EOF in infants with intestinal anastomosis.

**Methods** 568 infants from the multi-center cohort were divided into three types of intestinal anastomosis: duodenal anastomosis (EOF group,n=15; DOF group,n=67), jejunal anastomosis (EOF group,n=56;DOF group,n=155), and ileal/colonic anastomosis(EOF group,n=61;DOF group,n=214). The incidence of complications and the indexes of recovery were compared between the EOF and DOF groups in the three types of anastomosis independently.

Results Parenteral nutrition(PN) time and postoperative hospital stay were significantly shorter in EOF group than that in DOF group(Duodenal anastomosis:9.00[6.00,10.00] d vs 12.00[8.00,16.00] d,p=-0.033;10.00[7.00,13.00] d vs 14.00[11.00,18.00] d,p=0.002;Jejunal anastomosis:7.00[6.00,8.00] d vs 9.00[7.00,13.00] d,p<0.001;13.00[9.00,14.00] d vs 15.00[12.00,17.00] d,p<0.001;Ileal/colonic anastomosis:6.00[5.00,7.00] d vs 8.00[6.00,10.00] d,p<0.001;7.00[6.00,10.50] d vs 10.00[8.00,13.00] d,p<0.001). There were no differences in terms of abdominal distension,vomiting,diarrhea,weight change,serum albumin change,white blood cell(WBC) count,and C reaction protein(CRP) level at discharge between the EOF and DOF groups in the three types of anastomosis (all p>0.05). No hematochezia or anastomotic leakage were found.

#### Statistical analysis

Data were presented as percentages, medians, or averages, and the level of statistical significance was set at 0.05. SPSS 23.0 was used for statistical analysis, and the distribution of continuous variables was examined for normality. A t-test was applied for normally distributed data, and a rank-sum test was performed for non-normally distributed data. Categorical variables were tested using the chi-squared or Fisher's exact test.

**Results:**EOF in the three types of intestinal anastomosis in neonates and infants

| The types of intestinal | EOF | DOF | Chi-square test | |
|-------------------------|-------------|------------|-----------------|-------|
| anastomosis | [n(%)] | [n(%)] | χ2 | P |
| Duodenum(n=85) | 16(18.8%) | 69(81.2%) | | |
| Jejunum(n=211) | 60(28.2%) | 153(71.8%) | 6.657 | 0.036 |
| ileum/colon(n=275) | 68(19.3.2%) | 284(80.7%) | | |
| Total(n=568) | 144(23.2%) | 506(76.8) | - | - |

## Complications of EOF in the three types of intestinal anastomosis

| Complications | | Abdominal distension | vomit | diarrhea | overall<br>complication |
|---|---|---|---|---|---|
| | EOF(n=15) | 4(26.7%) | 4(26.7%) | 1(6.7%) | 7(46.7%) |
| Duodenal | DOF(n=67) | 13(19.4%) | 10(14.9%) | 3(4.5%) | 22(32.8%) |
| anastomosis | P | 0.501 | 0.275 | 0.562 | 0.375 |
| Jejunal<br>anastomosis | EOF(n=56) | 0(0.0%) | 4(7.1%) | - | 4(7.1%) |
| | DOF(n=155) | 8(5.2%) | 3(1.9%) | - | 11(7.1%) |
| | P | 0.113 | 0.082 | - | 1.000 |
| Ileal/Colonic anastomosis | EOF(n=61) | 4(6.6%) | 3(4.9% | 1(1.6% | 7(11.5%) |
| | DOF(n=214) | 6(2.8%) | 3(1.4%) | 2(0.9%) | 9(4.2%) |
| | p | 0.236 | 0.125 | 0.530 | 0.056 |

There were no hematochezia and anastomotic leakage in all types of intestinal anastomosis.

## Complications of EOF in the three types of intestinal anastomosis

| Compli | ications | Abdominal distension | vomit | diarrhea | overall<br>complication |
|---|---|---|---|---|---|
| D 1 1 | EOF(n=15) | 4(26.7%) | 4(26.7%) | 1(6.7%) | 7(46.7%) |
| Duodenal anastomosis DOF(n=6 | DOF(n=67) | 13(19.4%) | 10(14.9%) | 3(4.5%) | 22(32.8%) |
| | P | 0.501 | 0.275 | 0.562 | 0.375 |
| T ' 1 | EOF(n=56) | 0(0.0%) | 4(7.1%) | - | 4(7.1%) |
| Jejunal<br>anastomosis | DOF(n=155) | 8(5.2%) | 3(1.9%) | - | 11(7.1%) |
| | P | 0.113 | 0.082 | - | 1.000 |

| Ileal/Colonic anastomosis | EOF(n=61) | 4(6.6%) | 3(4.9% | 1(1.6% | 7(11.5%) |
|---|---|---|---|---|---|
| | DOF(n=214) | 6(2.8%) | 3(1.4%) | 2(0.9%) | 9(4.2%) |
| | p | 0.236 | 0.125 | 0.530 | 0.056 |

There were no hematochezia and anastomotic leakage in all types of intestinal anastomosis.

## **Study Design:**



# 2.The 2st part:Early oral feeding enhanced recovery after intestinal anastomosis in neonates and young infants less than 3 months old Abstract:

**Purpose** Early oral feeding(EOF) has been proven with a low incidence of complications and fast recovery after surgery in some elective pediatric patients, however, evidence for initiating EOF after intestinal anastomosis(IA) in neonates and young infants, with immature immune system and organs, is insufficient. This tudy was primary designed to investigate the status and evaluate the feasibility of EOF in neonates and young infants with IA in mainland china. **Method** 491 neonates and young infants from 51 hospital in china mainland were divided into two groups(EOF

group,n=88;traditional oral feeding,TOF group,n=403),and the clinical characteristics were collected and analyzed for evaluation of the status of EOF in neonates and young infants. The complications and recovery were also be compared to defined the feasibility after balancing the baseline by propensity score matching(PSM). Result The time of TPN,PN and postoperative hospital stay were significantly shorter in the EOF group than that in the TOF group in neonates and young infants with IA(2.00[1.00,2.00]d vs. 5.00[3.00,6.00]d, p<0.001; 7.00[5.00,8.00]d vs.9.00[7.00,13.00]d, p<0.001;11.00[8.00,14.00]]d vs.14.00[11.00,17.00]d). There were significant differences in the spectrum of disorders, anastomotic sites, operative age and weight between EOF and TOF groups(p=0.002;p=0.029,p=0.045,p<0.001). The overall low rate of EOF in neonates and infants with IA was 17.9%, especially lower in intestinal atresia, stenosis, stoma closure, ileal-colonic colonic anastomotic site operative age less than 30 days and weight less than 2.5kg. The overall rate of and Clavien-Dindo II complications were higher in EOF than TOF group(p=0.002),however,no differences were found complications(Clavien-Dindo III/ IV/V). Conclusion The rate of EOF in neonates and young infants with IA is low in Mainland China and the spectrum of disorders, an astomotic sites, operative age and weight maybe factors affecting the performing of EOF. Nevertheless, implementing EOF in neonates and young infants with IA maybe beneficial, enhances the recovery, and does not increase the rate of severe complications.

Keywords early oral feeding; intestinal anastomosis, neonate; young infant

#### Statistical analysis

Data were presented as percentages, medians, or averages, and the level of statistical significance was set at 0.05. SPSS 22.0 was used for statistical analysis, and the distribution of continuous variables was examined for normality. A t-test was applied for normally distributed data, and a rank-sum test was performed for non-normally distributed data. Categorical variables were tested using the chi-squared or Fisher's exact test. Before comparing the complications and recovery between EOF and TOF groups, a 1:2 propensity score match (PSM) with caliper 0.05 was applied to balance the baseline data between the two groups.

#### **Results:**

Baseline clinical characteristics of neonates and young infants with intestinal anastomosis in EOF and TOF groups

| group | | EOF | TOF | P |
|---|---|---|---|---|
| | | (n=88,%) | (n=403,%) | |
| The | Intestinal atresia(n=69) | 5 (5.7%) | 64 (15.9%) | 0.002 |
| spectrum | intestinal mass(n=32) | 4 (6.9%) | 28 (4.5%) | |
| of | intestinal necrosis(n=24) | 3 (5.2%) | 21 (3.4%) | |
| disorders | intestinal stenosis(n=38) | 3(3.4%) | 35(8.7%) | |
| | biliary disease(n=178) | 48(32.3%) | 130(54.5%) | |
| | colsing the stoma(n=41) | 4(4.5%) | 37(9.2%) | |
| | patent vitelline duct(n=19) | 6(n=3.2%) | 13(6.8%) | |
| | duodenal obstruction(n=84) | 15(17%) | 69(17.1%) | |
| | adhesional obstruction(n=6) | 0(0%) | 6(1.5%) | |
| Anastomic | Duodenal anastomosis | 15(17.0%) | 68(16.9%) | 0.029 |
| sites | (n=83) | | | |
| | Jejunal anastomosis(n=218) | 50(56.8%) | 168(41.7%) | |
| | Ileal anastomosis(n=123) | 19(21.6%) | 104(25.8%) | |
| | Ileal-colonic | 2(2.3%) | 34 (8.4%) | • |
| | anastomosis(n=36) | | | |
| | Colonic anastomosis(n=31) | 2(2.3%) | 29(7.2%) | |
| Surgical | laparoscope (n=132) | 19(21.6%) | 113(28.0%) | 0.216 |
| approach | laparotomy(n=359) | 69(78.4%) | 290(72.0%) | • |
| gender | male(n=259) | 46(52.37%) | 213(52.9%) | 0.921 |
| | female(n=232) | 42(47.7%) | 190(47.1%) | |
| Operative ag | ge (d,Median[P25%,P75%]) | 40[11,65] | 34[4,58] | 0.045 |
| ( | Operateive weight | 4.38[3.40,5.10] | 3.58[2.8,4.5] | < 0.00 |
| (kg,Median[P25%,P75%]) | | | | 1 |
| Pre-operative | | 37.10[34.63,40. | 36.30[33.10,39.7 | 0.054 |
| albumin(g | albumin(g/L,Median[P25%,P75%]) | | 0] | |
| | Pre-operative | 0.15[0.10,0.17] | 0.13[0.09,0.16] | 0.062 |
| prealbumin( | (g/L,Median[P25%,P75%]) | | | |

Baseline clinical characteristics of young infants with intestinal anastomosis in EOF and TOF groups after PSM

| | group | EOF | TOF | P |
|---|---|---|---|---|
| | | (n=86,%) | (n=156,%) | |
| The | Intestinal atresia(n=15) | 5(5.8%) | 11(7.1%) | 0.963 |
| spectrum | intestinal mass(n=15) | 4(4.7%) | 11(7.8%) | |
| of | intestinal necrosis(n=9) | 3(3.5%) | 6(3.8%) | |
| disorders | intestinal stenosis(n=11) | 3(3.5%) | 8(5.1%) | |
| | biliary disease(n=123) | 46(53.5%) | 77(49.4%) | |
| | colsing the stoma(n=13) | 4(4.7%) | 9(5.8%) | |
| | patent vitelline duct(n=13) | 6(n=7.0%) | 7(4.5%) | |
| | duodenal obstruction(n=42) | 15(17.4%) | 27(17.3%) | |
| Anastomic | Duodenal anastomosis | 15(17.4%) | 27(17.3%) | 0.927 |
| sites | (n=42) | | | |
| | Jejunal anastomosis(n=130) | 48(55.8%) | 82(52.6%) | |
| | Ileal anastomosis(n=60) | 19(22.1%) | 41(26.3%) | |
| | Ileal-colonic | 2(2.3%) | 2 (1.3%) | |
| | anastomosis(n=4) | | | |
| | Colonic anastomosis(n=6) | 2(2.3%) | 4(2.6%) | |
| Surgical | laparoscope (n=54) | 19(22.1%) | 35(22.4%) | 0.951 |
| approach | laparotomy(n=188) | 67(77.9%) | 121(77.6%) | |
| gender | male(n=130) | 44(51.2%) | 86(55.1%) | 0.554 |
| | female(n=112) | 42(48.8%) | 70(44.9%) | |
| Operative ag | ge (d,Median[P25%,P75%]) | 39.00[11.00,64. | 41.50[8.25,59.00 | 0.810 |
| | | 25] | ] | |
| Operateive weight | | 4.33[3.38,5.03] | 4.10[3.05,4.90] | 0.571 |
| (kg,N | Median[P25%,P75%]) | | | |
| | Pre-operative | 37.10[34.50,40. | 37.20[33.93,40.0 | 0.725 |

| albumin(g/L,Median[P25%,P75%]) | 15] | 0] | |
|---|---|---|---|
| Pre-operative | 0.15[0.11,0.17] | 0.14[0.10,0.17] | 0.515 |
| prealbumin(g/L,Median[P25%,P75%]) | | | |

# Recovery of young infants with intestinal anastomosis after EOF or TOF

| gruop | EOF(n=86) | TOF(n=156) | p |
|---|---|---|---|
| weight(kg,Median[P25%,P75%]) | 4.45[3.40,5.00] | 4.10[3.34,5.00] | 0.507 |
| albumin(g/L,Median[P25%,P75%]) | 36.73[34.00,41.50] | 37.15[34.23,41.48] | 0.510 |
| prealbumin(g/LMedian[P25%,P75%] | 0.15[0.11,0.19] | 0.14[0.11,0.18] | 0.255 |
| ) | | | |
| Time of | 2.00[1.00,2.00] | 5.00[3.00,6.00] | < 0.001 |
| TPN(d,Median[P25%,P75%]) | | | |
| Time of PN(d,Median[P25%,P75%]) | 7.00[5.00,8.00] | 9.00[7.00,13.00] | < 0.001 |
| Hospital | 11.00[8.00,14.00] | 14.00[11.00,17.00] | < 0.001 |
| stay(d,Median[P25%,P75%]) | | | |

## complications of young infants with intestinal anastomosis after EOF or TOF

| complications of young infants with intestinal anastomosis after Lot of Tor | | | | |
|---|---|---|---|---|
| gruop | | EOF | TOF(n=156,%) | p |
| | | (n=86,%) | | |
| Clavien-Dindo | Grade I (n,%) | 11(12.8%) | 14(9.0%) | 0.351 |
| classifification | Grade II(n,%) | 6(7.0%) | 0(0%) | 0.002 |
| | Grade III(n,%) | 0 | 1(0.6%) | 0.457 |
| | Grade IV/V(n,%) | 0 | 0 | - |
| | overall | 17 (19.8%) | 15 (9.6%) | 0.026 |
| Abdomir | nal distension | 12(14.0%) | 12(7.7%) | 0.119 |
| vomit | | 7(8.1%) | 1(0.6%) | 0.002 |
| diarrhea | | 1(1.2%) | 2(1.3%) | 0.936 |
| hematochezia | | 1(1.2%) | 0(0%) | 0.177 |
| anastom | otic leakage | 0(0%) | 1(0.6%) | 0.457 |

# Study design:

